CLINICAL TRIAL: NCT01668134
Title: Feasibility Study of Stereotactic Body Radiotherapy for Hepatocellular Carcinoma, and Intrahepatic Cholangiocarcinoma
Brief Title: Stereotactic Body Radiotherapy for Hepatocellular Carcinoma, and Intrahepatic Cholangiocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-1345 / 201107319
Record Dates: First submitted 2012-08-08; First posted 2012-08-17 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Carcinoma, Hepatocellular; Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stereotactic radiation (Experimental)
  Interventions: Radiation: Stereotactic radiation

INTERVENTIONS:
Radiation: Stereotactic radiation

SUMMARY:
This study is being done to determine if targeted radiation therapy (stereotactic) can be given to treat liver cancer, for patient who are unable to undergo surgery, over a short period of time with a small amount of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Karnofsky Performance Status of ≥ 60
* Pathologically confirmed IHC or HCC. (Pathology not required for HCC if the lesion enhances typically on MRI and the patient is evaluated by liver transplant surgery team and thought to have HCC.)
* 4 or less separate intrahepatic lesions, with at least one lesion that is able to be followed by EASL Criteria.
* Local surgical resection is not possible due to tumor or patient factors
* Limited metastatic disease is allowed if the volume of metastatic disease does not exceed the volume of primary disease.
* Prior TACE allowed if stopped/completed at least 2 weeks prior to enrollment
* Prior chemotherapy except Sorafenib allowed if stopped/completed at least 2 weeks prior to enrollment
* Prior Sorafenib allowed if stopped/completed at least seven days prior to enrollment.
* Able to provide signed informed consent

Exclusion Criteria:

* Childs-Pugh score 9 or more
* ALT or AST ≥ 6 x upper limit of normal
* Prior history of abdominal irradiation
* Women who are pregnant or nursing
* Scheduled to undergo chemotherapy except Sorafenib at the time when radiation therapy will be given, or for up to 4 weeks after completion of radiation therapy.
* Scheduled to undergo Sorafenib within seven days of when radiation therapy will be delivered, or for up to 2 weeks after completion of radiation therapy.
* Undergone prior radiation therapy to the abdomen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-12-16 (Actual); Primary Completion 2014-08-30 (Actual); Study Completion 2015-12-22 (Actual)

PRIMARY OUTCOMES:
Stereotactic radiation therapy (either photon or proton) can be delivered to the liver with a less than 10% 3-month incidence of Grade 4 study related toxicity. | Up to 90 days after end of radiation therapy

SECONDARY OUTCOMES:
Measure the late toxicity associated with using stereotactic radiation therapy in patients with unresectable HCC and IHC. | Up to 60 days after end of radiation therapy
Measure the local recurrence rates associated with using SBRT in patients with unresectable HCC and IHC. | Time of treatment until recurrance or progressive disease as measured by CT/MR from baseline to recurrance or progressive disease
Measure the overall survival rates associated with using SBRT in patients with unresectable HCC and IHC. | Baseline to time of death
Measure the response rates associated with using SBRT in patients with resectable HCC and IHC | Baseline to the first date of recurrance or progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: Parag Parikh, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu